CLINICAL TRIAL: NCT02787018
Title: Dexamethasone Compared With Dexmedetomidine as an Adjuvant to Ropivacaine for Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Parineeta Thapa, Dr, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRC/641/015
Record Dates: First submitted 2016-05-14; First posted 2016-06-01 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Brachial Plexus Block
Keywords: Brachial plexus block; Ropivacaine; Dexmedetomidine; Dexamethasone; Adjuvants, anesthesia
MeSH Terms: interventions — Ropivacaine; Saline Solution; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Block with Ropivacaine and Normal saline (Placebo Comparator): Patients will receive brachial plexus block with 20 ml 0.5% ropivacaine with 1ml normal saline: Total volume 21 ml
  Interventions: Drug: Ropivacaine and Normal saline
- Block with Ropivacaine and Dexamethasone (Active Comparator): Patients will receive brachial plexus block with 20ml 0.5% ropivacaine with 4mg (1ml) dexamethasone: Total volume 21 ml
  Interventions: Drug: Ropivacaine and Dexamethasone
- Block with Ropivacaine and Dexmedetomidine (Experimental): Patients will receive brachial plexus block with 20ml 0.5% ropivacaine with 50mcg (1ml) dexmedetomidine: Total volume 21 ml
  Interventions: Drug: Ropivacaine and Dexmedetomidine

INTERVENTIONS:
Drug: Ropivacaine and Normal saline — Supraclavicular brachial plexus block will be given with 0.5% ropivacaine with 1 ml normal saline
  Arms: Block with Ropivacaine and Normal saline
Drug: Ropivacaine and Dexamethasone — Supraclavicular brachial plexus block will be given with 0.5% ropivacaine with 4mg (1ml) dexamethasone
  Arms: Block with Ropivacaine and Dexamethasone
Drug: Ropivacaine and Dexmedetomidine — Supraclavicular brachial plexus block will be given with 0.5% ropivacaine with 50 mcg (1ml) dexmedetomidine
  Arms: Block with Ropivacaine and Dexmedetomidine

SUMMARY:
The investigators want to compare the effectiveness of dexamethasone and dexmedetomidine as an adjuvant to 0.5% ropivacaine for supraclavicular brachial plexus block on the onset of block and duration of analgesia, so that the investigators can choose the better adjuvant for the investigators routine practice of regional anesthesia.

DETAILED DESCRIPTION:
Ropivacaine is a newer local anesthetic which is structurally related to bupivacaine, but has fewer side effects. It is more cardio stable than bupivacaine, but the onset of action is delayed and the duration of action is shorter than bupivacaine making its use during regional anesthesia less preferable to many anesthesiologists. Steroids like dexamethasone, or alpha-2 agonists like dexmedetomidine are being studied as adjuvants to ropivacaine for brachial plexus block to improve its anesthetic properties and have shown favorable outcome in terms of shortening the onset of block and prolonging the duration of action. But no study has been done to compare their effects. So in this study the investigators want to compare the effectiveness of dexamethasone and dexmedetomidine as an adjuvant to 0.5% ropivacaine for supraclavicular brachial plexus block on the onset of block and duration of analgesia, so that the investigators can choose the better adjuvant for the investigators routine practice of regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists Physical Status I and II undergoing elective upper limb surgery under supraclavicular brachial plexus block

Exclusion Criteria:

* Patient's refusal to participate
* Patients weighing less than 40 kg
* Allergy to study drugs
* Infection at the site of injection
* Patients with preexisting neurological deficit
* Patients with diabetes mellitus
* Patients on steroids preoperatively
* Patients with bleeding disorder or coagulopathy
* Abnormalities in ECG like AV block or symptomatic bradycardia
* Patients receiving adrenoreceptor agonist or antagonist therapy preoperatively
* Requirement of conversion to general anesthesia due to inadequate block

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Onset of sensory block | every 3 minutes until 45 minutes after injection of drug
  Sensory block in the territories of median nerve (palmar surface of index finger), ulnar nerve (palmar surface of little finger), radial nerve (dorsal surface of first web space/ thumb) and musculocutaneous nerve (lateral side of volar surface of forearm) will be assessed by pinprick test using a 3-point scale:
  0 - normal sensation,
  1. - loss of sensation of pinprick (analgesia),
  2. - loss of sensation of touch (anaesthesia). Complete sensory block will be defined as grade 2 sensory block in 3 or more nerve territories.
Onset of motor block | every 3 minutes until 45 minutes after injection of drug
  Motor block will be evaluated by thumb flexion/ opposition (median nerve), thumb extension (radial nerve), finger abduction (ulnar nerve) and elbow flexion with forearm in full supination (musculocutaneous nerve) on a 3-point scale for motor function:
  0 - normal motor function,
  1. - reduced motor strength but able to move,
  2. - complete motor block. Complete motor block will be defined as grade 2 motor block in 3 or more nerve territories.
Duration of analgesia | Up to 24 hours after onset of block

SECONDARY OUTCOMES:
Duration of sensory block | Up to 24 hours after onset of block
  time from onset of sensory block to complete recovery of anaesthesia on all nerves.
Duration of motor block | Up to 24 hours after onset of block
  time from onset of motor block to the recovery of complete motor function of the hand and forearm
Incidence of side effects of drugs | Forty-eight hours following the injection of local anesthetics
  Side effects like bradycardia, tachycardia, hypotension, sedation, neurological deficit will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Parineeta Thapa, MD, Principal Investigator — BPKIHS, Dharan
Locations (1):
- B. P. Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Background] Das A, Majumdar S, Halder S, Chattopadhyay S, Pal S, Kundu R, Mandal SK, Chattopadhyay S. Effect of dexmedetomidine as adjuvant in ropivacaine-induced supraclavicular brachial plexus block: A prospective, double-blinded and randomized controlled study. Saudi J Anaesth. 2014 Nov;8(Suppl 1):S72-7. doi: 10.4103/1658-354X.144082. PMID 25538527 (Retraction: PMID 32934651 Saudi J Anaesth. 2020 Jul-Sep;14(3):422)
- [Background] Kumar S, Palaria U, Sinha AK, Punera DC, Pandey V. Comparative evaluation of ropivacaine and ropivacaine with dexamethasone in supraclavicular brachial plexus block for postoperative analgesia. Anesth Essays Res. 2014 May-Aug;8(2):202-8. doi: 10.4103/0259-1162.134506. PMID 25886227
- [Background] Zhang Y, Wang CS, Shi JH, Sun B, Liu SJ, Li P, Li EY. Perineural administration of dexmedetomidine in combination with ropivacaine prolongs axillary brachial plexus block. Int J Clin Exp Med. 2014 Mar 15;7(3):680-5. eCollection 2014. PMID 24753763